CLINICAL TRIAL: NCT05980897
Title: Inner Speech and Naming Treatment for Individuals with Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Mackenzie Fama, Assistant Professor, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCR224453
Record Dates: First submitted 2023-07-21; First posted 2023-08-08 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Aphasia; Anomia; Language Disorders; Communication Disorders
Keywords: Aphasia; Anomia; Speech-Language Pathology; Speech Therapy; Inner Speech
MeSH Terms: conditions — Aphasia; Anomia; Language Disorders; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Alternating treatment single-subject experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Naming Treatment (Experimental): Participants will complete three sessions of baseline probe testing (40 treatment items) occurring virtually on three consecutive days prior to treatment onset. Participants will then complete 10 sessions of therapy scheduled five days a week for two weeks, all occurring virtually. The treatment approach for this study will be a hierarchical, cueing-based treatment for naming.
  Interventions: Behavioral: Naming treatment

INTERVENTIONS:
Behavioral: Naming treatment — In this alternating treatment single-subject experimental design study, the investigators will alternate between two treatment conditions, i.e., two different types of stimulus items: those that are consistently reported as successful IS prior to treatment (sIS items) and those that are consistently reported as unsuccessful IS prior to treatment (uIS items). The treatment will be computerized to ensure consistency of presentation, timing, and cues across participants.
  For each stimulus presentation, the treatment hierarchy will proceed as follows:
  1. Name the picture independently
  2. Name the picture with a written cue
  3. Repeat the name of the picture
  4. Name the picture after a 5 second delay Each participant will be trained on a set of 40 items chosen specifically for them based on initial/baseline testing.

SUMMARY:
Aphasia is a language disorder, commonly resulting from stroke or other brain injury, that impacts a person's ability to communicate. This project is looking to improve upon current treatment methods for spoken naming in people with aphasia. People with aphasia frequently report being able to successfully say a word in their head, regardless of their ability to say the word out loud. For example, when presented with a picture of a house, they may report being able to think or hear "house" in their head, even if they can't name it out loud. This "little voice" inside one's head is known as inner speech (IS). Previous research suggests that some people with aphasia can re-learn to say words with successful IS (i.e., words they can already say in their heads) easier and faster than words with unsuccessful IS. This study will extend these findings by implementing a comparative treatment study in a larger group of participants with aphasia. The results will help to establish recommendations for speech-language pathologists in choosing treatment stimuli for anomia.

DETAILED DESCRIPTION:
Aphasia, a language disorder commonly acquired through stroke, has chronic negative impacts on communication abilities and quality of life. The specific language deficits associated with aphasia typically vary from person to person, but a universal element of aphasia is anomia, or difficulty with naming and word-finding. It is well-known that individuals with aphasia struggle to convey their ideas through overt speech, but little is known about this population's ability to access and utilize inner speech (IS). IS can be defined in many ways, but one simple definition that is well known to most language users is the mental imagery of having a little voice in one's head. Importantly, individuals with aphasia often endorse a mismatch between this "little voice" (IS) and what they can actually say out loud. In a prior interview-based study, over 75% of individuals with aphasia endorsed the specific experience of being able to say a word in their head despite being unable to say it aloud.

Previous research examined whether self-reported "successful IS" (sIS) (i.e., I can say the word in my head and it sounds right) predicted therapy outcomes in two participants. In both participants, self-reported IS predicted whether or not (and how quickly) individual words were successfully re-learned during a paired-associate treatment for anomia, and the effect was visible within just a few treatment sessions. This trial provides preliminary evidence that IS can be leveraged to improve outcomes of naming therapy for individuals with aphasia. This study aims to extend these prior finding by implementing a behavioral treatment for anomia using a single-subject experimental design in a larger group of individuals with aphasia.

The investigators predict that items reported as sIS will be more effectively learned during anomia treatment than items that are reported as uIS. Because sIS items are already being retrieved by the individual, one can think of them as being closer to successful spoken output than items that are not able to be retrieved (i.e., those reported as uIS).

ELIGIBILITY:
Inclusion Criteria:

* Have aphasia resulting from stroke occurring at least 6 months ago
* Are at least 18 years old
* Learned English at age 5 years or younger
* Normal or corrected-to-normal hearing and vision
* Have access to reliable internet at home for remote participation

Exclusion Criteria:

* Have a history of other brain conditions that could impact interpretation of results (such as Parkinson's Disease or dementia)
* Have a history of psychiatric disease requiring hospitalization, electroconvulsive therapy, or ongoing medication use (other than common antidepressants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Naming accuracy for sIS vs. uIS items (of 100%) | 5 weeks
  A direct comparison of treatment response for successful inner speech (sIS) vs. unsuccessful inner speech (uIS) items, measured via accuracy on a spoken naming test.

SECONDARY OUTCOMES:
Overall naming accuracy (of 100%) | 5 weeks
  A comparison of pre-treatment (average of three baseline sessions) to post-treatment spoken naming (40 items) across participants

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie Fama, Principal Investigator — The George Washington University
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data and/or testing materials with interested researchers, educators or clinicians upon request.
Time Frame: Data will be made accessible at the time of initial publication.
Access Criteria: Access to participant data by an external researcher may require a formal data sharing agreement with that researcher's institution.

REFERENCES:
- [Background] Fama ME, Hayward W, Snider SF, Friedman RB, Turkeltaub PE. Subjective experience of inner speech in aphasia: Preliminary behavioral relationships and neural correlates. Brain Lang. 2017 Jan;164:32-42. doi: 10.1016/j.bandl.2016.09.009. Epub 2016 Sep 29. PMID 27694017
- [Background] Fama ME, Snider SF, Henderson MP, Hayward W, Friedman RB, Turkeltaub PE. The Subjective Experience of Inner Speech in Aphasia Is a Meaningful Reflection of Lexical Retrieval. J Speech Lang Hear Res. 2019 Jan 30;62(1):106-122. doi: 10.1044/2018_JSLHR-L-18-0222. PMID 30950758
- [Background] Fama ME, Henderson MP, Snider SF, Hayward W, Friedman RB, Turkeltaub PE. Self-reported inner speech relates to phonological retrieval ability in people with aphasia. Conscious Cogn. 2019 May;71:18-29. doi: 10.1016/j.concog.2019.03.005. Epub 2019 Mar 25. PMID 30921682
- [Background] Fama ME, Turkeltaub PE. Inner Speech in Aphasia: Current Evidence, Clinical Implications, and Future Directions. Am J Speech Lang Pathol. 2020 Feb 21;29(1S):560-573. doi: 10.1044/2019_AJSLP-CAC48-18-0212. Epub 2019 Sep 13. PMID 31518502
- [Background] Hayward W, Snider SF, Luta G, Friedman RB, Turkeltaub PE. Objective support for subjective reports of successful inner speech in two people with aphasia. Cogn Neuropsychol. 2016 Jul-Sep;33(5-6):299-314. doi: 10.1080/02643294.2016.1192998. Epub 2016 Jul 29. PMID 27469037